CLINICAL TRIAL: NCT05069467
Title: Acupuncture Versus Sham Acupuncture or Usual Care for Antiandrogen-Induced Hot fLashes in Prostate Cancer (AVAIL): a Multicenter Randomized Controlled Trial
Brief Title: Acupuncture Versus Sham Acupuncture or Usual Care for Antiandrogen-Induced Hot fLashes in Prostate Cancer (AVAIL)
Acronym: AVAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: West China Hospital (Other); Yantai Hospital of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Jiani Wu, Dr., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020030KY02
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hot Flashes; Prostate Cancer; Acupuncture
Keywords: Prostate Cancer; Hot Flashes; Acupuncture; Randomized Controlled Trial
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly 2:1:1 allocated to the verum acupuncture (n=60), sham acupuncture (n=30), or usual care (n=30) group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The principal investigator, study investigators, patients, study staff, and the statistician will be blinded to the treatment assignments among interventions. The acupuncturists cannot be blinded to verum acupuncture or the sham owing to the characteristics of acupuncture procedure. Patients allocated to both verum acupuncture and sham acupuncture groups will be asked to guess which type of acupuncture (verum acupuncture, sham acupuncture, or unclear) they had received after the end of last treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture (Experimental): Licensed acupuncturists with more than 5 years of experience will be responsible for administering interventions three times per week for 6 weeks. The needles (30 or 40 mm and 0.25 mm gauge; Soochow, Hwato) will be inserted and manipulated until De Qi, a sensation of soreness and tingling. Acupuncture was defined as targeting the 10 bilateral acupuncture points: Xinshu (BL15), Shenshu (BL23), Zhongliao (BL33), Sanyinjiao (SP6), Yinlingquan (SP9). The needle will be left in place for 30 minutes with brief manipulation at the beginning, middle, and end of therapy.
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Treatment will be the same for the sham acupuncture, except for the following: the acupuncturist selected the same number of nonacupuncture, nontrigger points. Instead of eliciting De Qi, the needles will be minimally manipulated to avoid eliciting sensations other than initial contact with skin.
  Interventions: Device: Sham Acupuncture
- Usual Care (No Intervention): Patients receiving usual care received neither acupuncture nor sham acupuncture. After the 6-week assessment, patients will be offered the option to receive acupuncture treatment as the acupuncture group.

INTERVENTIONS:
Device: Acupuncture — For the active acupuncture group, the acupuncturist chose standard points depending on subjects' preferred positions. In addition, up to four acupuncture points were chosen on the basis of subjects' other presenting symptoms (such as fatigue, insomnia, or erectile dysfunction). The needles (30 or 40 mm and 0.25 mm gauge; Soochow, Hwato) will be inserted and manipulated until De Qi, a sensation of soreness and tingling.
  Arms: Acupuncture
Device: Sham Acupuncture — Treatment will be the same for the sham acupuncture, except for the following: the acupuncturist selected the same number of nonacupuncture, nontrigger points. Instead of eliciting De Qi, the needles will be minimally manipulated to avoid eliciting sensations other than initial contact with skin.
  Other Names: Placebo Needle; Non-penetrating Acupuncture
  Arms: Sham Acupuncture

SUMMARY:
Hot flashes are a common and debilitating symptom among prostate cancer patients undergoing androgen deprivation therapy (ADT). Strong evidence from multiple rigorously designed studies indicated that venlafaxine provides partial relief, but the tolerability is poor when the dose is not tapered. Hence, an alternative therapy is needed. Previous studies reported that acupuncture may be helpful in the management of hot flashes. However, the insufficient randomized controlled trial limited the quality of evidence.

DETAILED DESCRIPTION:
The number of men surviving after being diagnosed with prostate cancer has increased rapidly. According to population-based cancer registry data, 10-year survival has tripled in the past 40 years in the UK. Androgen deprivation therapy (ADT) is a mainstay of prostate cancer treatment and has been shown in randomized controlled trials to improve overall survival when used with radiation for intermediate- and high-risk localized disease, as well as locally advanced and node-positive disease, and after surgery for the node-positive disease. Although ADT can improve survival, it can also cause significant morbidity and a decrement in quality of life. One of the most bothersome side effects is hot flashes. They are experienced as sudden and transient episodes of heat and sweating, with possible co-occurring palpitations and anxiety, usually persist long-term. The prevalence estimated that 44-80% of patients undergoing ADT report hot flashes and up to 27% report this as the most troublesome adverse effect. Although hot flashes are not fatal morbidity, it may interfere with adherence to lifesaving therapies or ablative therapies that are used to prevent or treat cancer.

Currently, most intervention studies for hot flashes have evaluated treatments in breast cancer patients or women who are postmenopausal. Venlafaxine, a selective serotonin reuptake inhibitor, appears to be effective and safe in both breast cancer women and prostate cancer men with hot flashes. It has been recommended for practice in men with strong evidence from multiple rigorously designed studies. However, some prostate cancer patients cannot take venlafaxine because of side effects such as nausea, headache, dry mouth, dizziness, insomnia, and constipation. Thus, an alternative therapy is needed. A systematic review identified six studies of acupuncture for hot flashes, of which none were randomized and placebo-controlled. Although acupuncture is a nonpharmacologic therapy and has been confirmed that could be helpful in the management of hot flashes among breast cancer survivors, there is no placebo acupuncture-controlled trials demonstrating its efficacy in men.

ELIGIBILITY:
Inclusion Criteria:

* patients aging from 18 to 75 years diagnosed with prostate cancer undergoing ADT;
* with an average of 3 or more hot flashes a day for at least 3 days before enrollment and no other clinically significant disease;
* not receiving any medications for hot flashes nor did they have a previous history of acupuncture treatment.

Exclusion Criteria:

* hormonal treatment other than GnRH analogue
* daily treatment with psychotropic drugs
* newly started or changed alternative medications with possible effects on flushes uncontrolled hypertension or metabolic disease
* inability to move/lie on the side, and treatment with anticoagulants or pacemaker.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Weekly mean hot flash symptom severity score (HFSSS) | Baseline to week 6
  The HFSSS is defined as the product of "hot frequency" and "hot severity". The severity of hot flashes is assessed based on the duration of hot flashes and physical and emotional symptoms; it is scored as mild, moderate, severe, and very severe (range 1-4, from mild to very severe).

SECONDARY OUTCOMES:
Weekly mean hot flash symptom severity score (HFSSS) | Baseline to week 14
  The HFSSS is defined as the product of "hot frequency" and "hot severity". The severity of hot flashes is assessed based on the duration of hot flashes and physical and emotional symptoms; it is scored as mild, moderate, severe, and very severe (range 1-4, from mild to very severe).
Response rate of HFSSS | Baseline, week 6, and week 14
  The responders will be defined according to a 50% reduction of HFSSS
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | Baseline, week 6, and week 14
  The Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire is a relevant, worldwide tool used for assessing the health-related quality of life in men with prostate cancer.
International Index of Erectile Function (IIEF-5) | Baseline, week 6, and week 14
  The IIEF-15 comprises 15 items divided into 5 domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction, respectively. The IIEF-5 comprises 5 items from the IIEF-15, 4 from the erectile function domain, and 1 from intercourse satisfaction. Response options for each item ranged from 1 to 5, and occasionally the option "0" depicting no sexual stimulation/intercourse, the scores are summed.
The Zung Self-Rating Anxiety Scale (SAS) | Baseline, week 6, and week 14
  The SAS consists of 20 items that assess common symptoms of anxiety, such as tension, fear, worry, and nervousness. Each item is rated on a Likert-type scale ranging from 1 to 4. Scores on the scale can rage from 20 to 80, with higher scores indicating more severe symptoms of anxiety.
The Zung Self-Rating Depression Scale (SDS) | Baseline, week 6, and week 14
  The SDS is a 20-item measure, with each item rated on a 4-point scale. It requires approximately 5-10 minutes to complete. Ranges for mild to moderate depression, moderate to severe depression, and severe depression are 50-59, 60-69, and over 70, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jiani Wu, M.D., Ph.D., Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Jiangsu Cancer Hospital & Jiangsu Institute of Cancer Research & Nanjing Medical University Affiliated Cancer Hospital, Nanjing, Jiangsu
  - Yantai Hospital of Traditional Chinese Medicine, Yantai, Shandong
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
The deidentified participant data will be shared after publication. Researchers can access the data with a specific purpose and a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: With publication
Access Criteria: For a specified purpose with a signed data access agreement

REFERENCES:
- [Derived] Qin Z, Zang Z, Yu J, Lv J, Li N, Zhang J, Yang M, Kwong JSW, Pang R, Wang J, Cui Z, Yu Y, Wang H, Zhu Y, Yuan Y, Li X, Wu Y, Wu J. Acupuncture versus sham acupuncture and usual care for Antiandrogen-Induced hot fLashes in prostate cancer (AVAIL): study protocol for a randomized clinical trial. BMC Complement Med Ther. 2023 Oct 27;23(1):388. doi: 10.1186/s12906-023-04218-y. PMID 37891531